CLINICAL TRIAL: NCT07231549
Title: CuidAME: Longitudinal Data Collection From Patients With Spinal Muscular Atrophy in Spain
Acronym: CUIDAME
Status: Recruiting | Type: Observational
Sponsor: Fundació Sant Joan de Déu (Other)
Responsible Party: Sponsor
Other Study IDs: EOM-24-02
Record Dates: First submitted 2025-06-17; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-02

CONDITIONS: Spinal Muscular Atrophy
Keywords: registry; natural history; adult; pediatric
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Subjects with Spinal Muscular Atrophy 5q: Subjects with Spinal Muscular Atrophy 5q

SUMMARY:
The goal of this observational study is to set up a longitudinal data collection study to perform a long-term follow-up of SMA patients in a real-world setting, and to standardise and homogenize the data collection process for SMA patient's data.

Treated and untreated patients will be followed based on the routine clinical practice schedule.

DETAILED DESCRIPTION:
This is a retrospective, prospective, multicentre, non-randomized data collection study in Spain. The dataset collected is based on the TREAT-NMD SMA Core Dataset and the CuidAME steering committee consensus. The study collects pseudo-anonymized data, including data on genetic test results, clinical diagnoses, treatment, and outcome measures.

Patients will be followed based on the routine clinical practice schedule. Motor outcomes will be captured regularly, following the SMA standards of for care, for patients with a DMT every 6 months or at least once per year in patients without DMTs, for at least a 5-year follow-up period initially, which could be extended under agreement with funders of the study.

Participation in this study does not modify or influence any clinical decisions regarding the treatment the patient may receive, clinical assessments performed or frequency of visits.

The study will not collect data from patients participating in a clinical trial from the time they are enrolled. Data collected before the enrolment may be used, and data collection may continue after the end of the clinical trial. Data generated during a clinical trial could be used if written permission from the clinical trial sponsor is obtained.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed 5q SMA
* Patient or caregivers written informed consent has been obtained (except for paediatric patients deceased).

Exclusion Criteria:

* Further types of SMA (non-5q SMA).
* Patient without legal capacity who cannot understand the nature, significance, and consequences of the project.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will collect data from SMA patients in Spain, independently of their treatment regimen, age, or disease status, from April 2020 onwards.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-05-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Motor and functional status (WHO) | Yearly through study completion, an average of 5 years
  Motor status will be captured (all patients): WHO motor milestones: checklist that assesses whether a child can sit independently, crawl, stand with/without support, and walk with/without support. Changes in this score (loss or gain in function) and maintenance of score throughout study duration is assessed.
Motor and functional status (CHOP INTEND) | Yearly through study completion, an average of 5 years
  Motor status will be captured (patients below two years of age): Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP INTEND): maximum score of 64.
Motor and functional status (HFMSE) | Yearly through study completion, an average of 5 years
  Motor status will be captured (patients over 36 months of age): Hammersmith Functional Motor Scale Expanded (HFMSE): maximum score of 66.
Motor and functional status (RULM) | Yearly through study completion, an average of 5 years
  Motor status will be captured (patients obver 36 months of age): Revised Upper Limb Module (RULM): maximum score of 37.
Motor and functional status (6MWT) | Yearly through study completion, an average of 5 years
  Motor status will be captured (ambulant patients): 6-Minute-Walk Test (6MWT): walked distance within 6 min.

SECONDARY OUTCOMES:
Clinical SMA characteristics: mechanical ventilation | Through study completion, an average of 5 years
  Change in mechanical ventilation prevalence: percent of participants who required ventilatory support (invasive or non-invasive)
Clinical SMA characteristics: external nutrition | Yearly through study completion, an average of 5 years
  Change in external nutrition prevalence: percent of participants who required external nutrition support
Clinical SMA characteristics: scoliosis | Yearly through study completion, an average of 5 years
  Change in scoliosis presence or scoliosis surgery prevalence: percent of participants who presented scoliosis and percent of participants with spinal surgery.
Clinical SMA characteristics: neurodevelopmental developoment | Yearly through study completion, an average of 5 years
  Prevalence of neurodevelopmental disorders: percentage of patients who, after assessment by a neuropaediatrician, present with language, behavior, social or understanding alterations
Clinical SMA characteristics: treatment sequence | Yearly through study completion, an average of 5 years
  change in treatments: distribution of patients in the different possible treatment sequences

CONTACTS AND LOCATIONS:
Overall Officials: Andrés Nascimento, Study Chair — Hospital Sant Joan de Deu; Mónica Povedano Panadés, Study Chair — Hospital Universitari de Bellvitge; Francina Munell Casadesús, Study Chair — Hospital Universitari Vall d'Hebrón; Miguel Angel Fernández García Miguel Angel Fernández García, Study Chair — Hospital Universitario La Paz; Inmaculada Pitarch Castellano, Study Chair — Hospital Universitario La Fe; Juan Francisco Vázquez Costa, Study Chair — Hospital Universitario La Fe; Maria Grazia Cattinari, Study Chair — Fundación Atrofia Muscular Espinal; Rocío Calvo, Study Chair — Hospital Universitario Regional de Málaga; Eduardo Martínez Salcedo, Study Chair — Hospital Universitario Virgen de la Arrixaca; Antonio Moreno Escribano, Study Chair — Hospital Universitario Virgen de la Arrixaca; Julita Medina Cantillo, Study Chair — Hospital Sant Joan de Deu
Locations (1):
- Hospital Sant Joan de Déu, Esplugues de Llobregat, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.registro-cuidame.org/